CLINICAL TRIAL: NCT05321108
Title: Aerobic Exercise Versus Whole-Body Vibration On Fatigue, Functional Capacity And Quality Of Life In Patients With Systemic Lupus Erythematosus: A Randomized Controlled Trial
Brief Title: Aerobic Exercise Versus Whole-Body Vibration on Fatigue, Functional Capacity, Quality of Life in Systemic Lupus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ereny Sobhy Wahba Khalil, Assistant professor of physical therapy for surgery - Faculty of physical therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003502
Record Dates: First submitted 2022-03-06; First posted 2022-04-11 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Systemic; Lupus
Keywords: Aerobic; Exercise; Systemic; Lupus; Whole; Body; Vibration
MeSH Terms: conditions — Motor Activity | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Procedures of the study:
  The assessment procedures
  1. Measuring of functional capacity and health-related quality of life in Systemic Lupus by: The Systemic Lupus Erythematosus Quality of Life (SLEQOL) questionnaire (Arabic version of the SLEQOL) 2- Measuring of functional capacity in Systemic Lupus by: Health Assessment Questionnaire (HAQ) The Arabic- Health Assessment Questionnaire (HAQ) 3- Measuring of fatigue in Systemic Lupus by: Fatigue severity scale (Arabic version of the FSS-Arabic) (FSS-Ar):
  Therapeutic procedures:
  1. Aerobic exercise
  2. Whole-body vibration (WBV)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (GA) (Aerobic exercise group): (Experimental): the patient will receive aerobic exercise program: (graded treadmill machine walking and stepping exercises). The second part of the exercise program will be 10 minutes of stepping exercise at a speed of 96 beats per minute using a 20-cm-high bench, with rest after the first 5 minutes. Three sessions per week for 12 weeks.
  Interventions: Other: Group B (GB) (Whole-body vibration (WBV) group)
- Group B (GB) (Whole-body vibration (WBV) group) (Experimental): the patient will receive whole-body vibration with frequency 30-40Hz and 2 mm of amplitude will be used for the whole-body vibration program by reciprocating vertical displacements on the left and right side of a fulcrum. The WBV group performed a training program 3 times a week with at least one day between each session for 12 weeks.
  Interventions: Other: Group A (GA)(Aerobic exercise group)

INTERVENTIONS:
Other: Group A (GA)(Aerobic exercise group) — Aerobic Exercise has been demonstrated to be a safe strategy to improve several health outcomes in Systemic lupus erythematosus (SLE)SLE, including depressive symptoms or, even more importantly, fatigue and quality of life.
  Arms: Group B (GB) (Whole-body vibration (WBV) group)
Other: Group B (GB) (Whole-body vibration (WBV) group) — (WBV) has been growing over the years. WBVE occurs when the subject is in contact with the vibrating platform in operation and is exposed to the generated mechanical vibrations. WBV has a positive action on muscle strength, bone formation, balance, flexibility, functional capacity and fatigue.
  Arms: Group A (GA) (Aerobic exercise group):

SUMMARY:
PURPOSE: … The aim of this study will be conducted to investigate the therapeutic efficacy of Aerobic exercise versus whole-body vibration on fatigue, functional capacity and quality of life in patients with systemic lupus erythematosus

RESEARCH QUESTION:

The problem of the study will be designed in a questioner form " which is more effective Aerobic Exercise or Whole-Body Vibration on Fatigue, Functional Capacity And Quality Of Life In Patients With Systemic Lupus Erythematosus?

DETAILED DESCRIPTION:
Procedures of the study:

The assessment procedures

1. Measuring of functional capacity and health-related quality of life in Systemic Lupus Erythematosus patients by:

   The Systemic Lupus Erythematosus Quality of Life (SLEQOL) questionnaire SLEQoL is a 40-item questionnaire that was developed and validated in an English-speaking cohort of SLE patients in Singapore and it assesses the quality of life of Systemic Lupus Erythematosus (SLE) patients across six domains including physical functioning, occupational activities, symptoms, treatment, mood and self-image.

   Arabic version of the SLEQOL The questionnaire which is a reliable and valid specific instrument for measuring the quality of life of Egyptian SLE patients, cross-cultural adaptation and validation of SLEQoL has been performed in Arabic (Egypt). Each domain score varies from 1 to 7, with higher scores indicating poorer quality of life. The total scores of the questionnaire vary between 40 and 280.

   The Arabic version of the SLEQOL is used to measure health-related quality of life in Systemic Lupus Erythematosus patients pre-treatment (pre-test) and after 6 weeks (post-treatment 1) and after 12 weeks of the study (post-treatment 2).
2. Measuring of functional capacity in Systemic Lupus Erythematosus patients by:

   Health Assessment Questionnaire(HAQ)

   HAQ has been reported as the best tool targeting functional disability. Moreover, the validity and reliability of the HAQ have been confirmed in several ethnic groups. It contains 20 questions grouped into eight subscales (dressing and grooming, arising, eating, walking, hygiene, reach, grip, activities). The response categories are "without any difficulty" (score = 0),"with some difficulty" (score = 1), "with much difficulty" (score = 2), and "unable to do" (score = 3). The highest score for any question determines the score for the subscale in question. The use of any assistive device or any other person's help was given a score of 2. The HAQ disability index was calculated as the sum of the scores for various subscales, divided by the number of subscales responded to, and results in a score between 0 and 3.

   The Arabic- Health Assessment Questionnaire(HAQ) The Arabic HAQ is a reliable and valid instrument that can be self-administered to Arabic patients to evaluate their functional disability.

   The Arabic HAQ is used to measure functional capacity in Systemic Lupus Erythematosus patients pre-treatment (pre-test) and after 6 weeks (post-treatment 1) and after 12 weeks of the study (post-treatment 2).
3. Measuring of fatigue in Systemic Lupus Erythematosus patients by:

Fatigue severity scale The Fatigue severity scale (FSS) is a self-reported questionnaire It consists of 9 statements that rate the severity of the patient's fatigue symptoms in terms of how these symptoms affect motivation, exercise, physical function, and activities of daily living. Reflecting on their condition, patients score each item from 1 to 7, based on the extent, to which they agree or disagree with each statement (1 = strong disagreement, 7 = strong agreement). The FSS can be scored either by obtaining a total score or by calculating a mean score across all 9 items, with higher scores indicating more severe fatigue. The most appropriate tool to measure fatigue in SLE. The FSS is widely used in clinical practice and research and has been translated into several languages.

Arabic version of the FSS-Arabic (FSS-Ar) The development of an Arabic version of the FSS-Arabic (FSS-Ar) and its validation would be of great value, as it would allow clinicians and researchers to investigate the incidence and impact of fatigue associated with it.

The Arabic version of the FSS-Arabic (FSS-Ar) is used to measure fatigue in Systemic Lupus Erythematosus patients pre-treatment (pre-test) and after 6 weeks (post-treatment 1) and after 12 weeks of the study (post-treatment 2).

Therapeutic procedures:

This current study will be designed to determine which is more effective aerobic exercise or whole-body vibration on fatigue, functional capacity and quality of life in patients with systemic lupus erythematosus so the treatment protocol will be applied through the following steps and phases:

Therapeutic intervention for the study will be started at the same time for all groups of the study as follows;

1. Aerobic exercise

   Exercise Program:
   * The program will consist of three 50-minute exercise sessions weekly over 12 weeks.
   * Each exercise session included graded treadmill machine walking and stepping exercises. Maximal exercise tolerance test (Bruce protocol) will be performed on the preceding day of the exercise program. Maximum heart rate is calculated by the formula (220 -age).
   * The graded treadmill machine walking exercise will be started with a 5-minute warm-up period with the intensity of about 40% of maximum heart rate followed by a 30-minutes training phase. The training intensity will be arranged at about 70-85% of maximum heart rate and ended with a 5-minute cool-down period with the intensity of about 40% of maximum heart rate. Exercising sessions will be comprised of warming up (stretching, turning joints, and walking slowly), the main program (treadmill machine walking), and cooling down (stretching, turning joints, and walking slowly).
   * The second part of the exercise program will be 10 minutes of stepping exercise at a speed of 96 beats per minute using a 20-cm-high bench, with rest after the first 5 minutes.
2. Whole-body vibration (WBV)

   * Whole-body vibration apparatus (model power plate-my5tm, made in the United States) with frequency 30-40Hz and 2 mm of amplitude will be used for whole-body vibration program by reciprocating vertical displacements on the left and right side of a fulcrum.
   * The subjects will stand on a whole-body vibrator and they will be vibrated in a squat positioning.
   * The subjects will exercise for 16 minutes (1 min vibration with 8 iterations and 1 min break between each iteration), 20, and 24 minutes in the first week to the third week, the fourth week to the sixth week, and the seventh week to the eighth week respectively and also to the end of the study after 12 weeks.
   * The WBV group performed a training program 3 times a week with at least one day between each session for 12 weeks.

Treatment procedure Interventions

Participants were randomly assigned to:

* Group A (GA) (Aerobic exercise group): Will receive aerobic exercise: (graded treadmill machine walking and stepping exercises). The second part of the exercise program will be 10 minutes of stepping exercise at a speed of 96 beats per minute using a 20-cm-high bench, with rest after the first 5 minutes. Three sessions per week for 12 weeks.
* Group B (GB) (Whole-body vibration (WBV) group): will receive whole-body vibration with frequency 30-40Hz and 2 mm of amplitude will be used for the whole-body vibration program by reciprocating vertical displacements on the left and right side of a fulcrum. The WBV group performed a training program 3 times a week with at least one day between each session for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for selecting the patients include the following:

  * This study turned will be done on 68 patients.
  * Age range between 25-45 years.
  * Female patients with a diagnosis of Systemic Lupus Erythematosus (SLE).
  * A follow-up of 12 months.
  * Clinical and treatment stability during the 6 previous months.
  * Not performing regular exercise.
  * All patients enrolled in the study will have their informed consent

Exclusion Criteria:

* The subjects are excluded from the study if they will meet one of the following criteria;

  * Have had biological treatment in the previous 6 months.
  * A background of clinical cardiovascular disease in the previous year.
  * Present contraindications to performing the exercise.
  * Other associated rheumatic diseases, pregnancy, active acute or chronic infection.
  * Acute renal failure, cardiac or pulmonary involvement.
  * Have a depressive disorder.
  * Undergo total hip replacement.
  * Diabetes, cancer.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Health Assessment Questionnaire(HAQ) | 2 hours
  Health Assessment Questionnaire (HAQ)It contains 20 questions grouped into eight subscales The response categories are "without any difficulty" (score = 0),"with some difficulty" (score = 1), "with much difficulty" (score = 2), and "unable to do" (score = 3).
Measuring of fatigue in Systemic Lupus Erythematosus patients by: Fatigue severity scale | 2 hours
  Fatigue severity scale The Fatigue severity scale (FSS) is a self-reported questionnaire It consists of 9 statements that rate the severity of the patient's fatigue symptoms in terms of how these symptoms affect motivation, exercise, physical function, and activities of daily living. Reflecting on their condition, patients score each item from 1 to 7, based on the extent, to which they agree or disagree with each statement (1 = strong disagreement, 7 = strong agreement).
  Arabic version of the FSS-Arabic (FSS-Ar) The development of an Arabic version of the FSS-Arabic (FSS-Ar) and its validation would be of great value, as it would allow clinicians and researchers to investigate the incidence and impact of fatigue associated with it
functional capacity and health-related quality of life The Systemic Lupus Erythematosus Quality of Life (SLEQOL) questionnaire | 2 hours
  SLEQoL is a 40-item questionnaire and it assesses the quality of life of Systemic Lupus Erythematosus (SLE) patients across six domains including physical functioning, occupational activities, symptoms, treatment, mood and self-image. Each domain score varies from 1 to 7, with higher scores indicating poorer quality of life. The total scores of the questionnaire vary between 40 and 280.

CONTACTS AND LOCATIONS:
Overall Officials: Ereny S. Wahba khalil, Asst.Prof.Dr, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy. Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No